CLINICAL TRIAL: NCT00087451
Title: A Phase I Sequential Ascending Dose Trial of AP23573 in Patients With Progressive or Recurrent Malignant Glioma
Brief Title: Safety Study of AP23573 in Patients With Progressive or Recurrent Glioma (8669-023)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-023; AP23573-04-103
Record Dates: First submitted 2004-07-08; First posted 2004-07-13 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Malignant Glioma; Glioblastoma; Gliosarcoma
Keywords: Progressive or recurrent malignant glioma
MeSH Terms: conditions — Glioma; Glioblastoma; Gliosarcoma | interventions — ridaforolimus

INTERVENTIONS:
Drug: AP23573 — ridaforolimus
  Other Names: deforolimus; MK-8669; ridaforolimus was also known as deforolimus until May 2009

SUMMARY:
A Phase I, open-label, non-randomized, sequential dose escalation cohort trial of the safety, tolerability, and maximum tolerated dose (MTD) of AP23573 when administered intravenously as a 30-minute infusion, once daily for five days, repeated every two weeks, to patients with progressive or recurrent malignant glioma.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the safety, tolerability, and maximum tolerated dose (MTD) of AP23573 when administered intravenously once daily for five days repeated every two weeks to patients with progressive or recurrent gliomas who have failed standard therapy and who are or are not receiving enzyme-inducing anticonvulsant (EIAC) medications.

The secondary objectives are to: characterize the pharmacokinetic profile of AP23573 when administered daily for five days repeated every two weeks at the indicated dosage levels in patients receiving and not receiving EIAC; describe the progression-free survival at six months; describe changes in proteins affected by mTOR inhibition; describe single timepoint status of proteins affected by mTOR inhibition in tumor tissue surgical specimens after AP23573 dosing; describe the status of key proteins in the mTOR signaling pathway in archival tumor samples, if available; describe health-related quality of life at the start of the trial and prior to study drug infusion and at various timepoints throughout the trial.

Protocol Outline:

This is a Phase I, open-label, non-randomized, sequential dose escalation cohort trial of the safety, tolerability, and MTD of AP23573 when administered intravenously as a 30-minute infusion, once daily for five days, repeated every two weeks, to patients with progressive or recurrent malignant glioma.

ELIGIBILITY:
Inclusion Criteria (Patients must meet each of the following criteria to be eligible for participation in the trial):

* Male or female patients ≥ 18 years of age
* Patients must have a radiographically suspected progressive or recurrent primary malignant glioma (glioblastoma multiforme or gliosarcoma) and must have failed standard therapy. Patients may not have received any systemic therapy for the treatment of this recurrence or relapse
* Patients must be candidates for surgical resection or open biopsy of the tumor
* Patients who have had previous surgical resection(s) are eligible
* Patients must have had minimum prior therapy of radiotherapy and documented progression of disease thereafter
* Patients must have had a tissue proven malignant glioma
* A minimum interval of at least four weeks prior to the first dose of AP23573 must have elapsed for all patients enrolling after either prior surgery or completion of prior external beam radiotherapy for initial primary diagnosis
* A minimum interval of four weeks prior to the first dose of AP23573 must have elapsed since receipt of any investigational therapy or any other chemotherapy
* Patients in the EIAC cohorts must be presently receiving a stable dose of EIAC (e.g., dilantin, phenytoin, etc.) for at least two weeks prior to the first dose of AP23573
* For patients on corticosteroids, the dose must be stable for at least one week prior to the first dose of AP23573
* Patients must be neurologically stable for at least two weeks prior to the first dose of AP23573
* Patients must have an ECOG performance status of 0 or 1
* Patients must either not be of childbearing potential or have agreed to use a medically effective method of contraception
* Patients must have adequate hematologic, renal and liver function as specified in the protocol
* Patients must be able to understand and give written informed consent

Exclusion Criteria (Patients meeting any of the following criteria are ineligible for participation in the trial):

* Women who are pregnant or lactating
* Patients with known or suspected hypersensitivity to either drugs formulated with polysorbate 80 (Tween) or any other excipient contained in the study drug formulation
* Patients with known hypersensitivity to macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin)
* Patients with significant cardiovascular disease, as specified in the protocol
* Patients with known HIV infection
* Patients with any active infection requiring prescribed intervention
* Patients receiving immunosuppressive agents other than prescribed corticosteroids
* Patients who have had prior therapy with rapamycin, any rapamycin analog or tacrolimus
* Patients with inadequate recovery from any prior surgical procedure or patients having undergone any major surgical procedure within two weeks prior to the first dose of AP23573
* Patients with any other life-threatening illness or organ system dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with evaluation of the safety of the study drug
* Patients with a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies
* Patients with another primary malignancy within the past three years (except for non-melanoma skin cancers and cervical carcinomas in situ)
* Patients with the inability, in the opinion of the Investigator, to comply with the protocol requirements
* Patients are not permitted any chemotherapeutic agents or other antineoplastic agents either during or within four weeks prior to the first dose of AP23573. Additional excluded drugs and treatments are specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Center For Neuro-Oncology, Dana Farber Cancer Institute, Boston, Massachusetts
  - The Brain Tumor Center at Duke, Duke University Medical Center, Durham, North Carolina
  - Brain Tumor Institute, The Cleveland Clinic, Cleveland, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Reardon DA, Wen PY, Alfred Yung WK, Berk L, Narasimhan N, Turner CD, Clackson T, Rivera VM, Vogelbaum MA. Ridaforolimus for patients with progressive or recurrent malignant glioma: a perisurgical, sequential, ascending-dose trial. Cancer Chemother Pharmacol. 2012 Apr;69(4):849-60. doi: 10.1007/s00280-011-1773-y. Epub 2011 Oct 30. PMID 22037923